CLINICAL TRIAL: NCT02159378
Title: Fructosamines and Gestational Diabetes (FRUCTO)
Acronym: FRUCTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHD008-14
Record Dates: First submitted 2014-06-06; First posted 2014-06-09 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy; Gestational Diabetes
Keywords: Gestational Diabetes; Fructosamines; Insulin treatment
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GD with Insulin treatment (Other): At the end of the study patients will be divided into two groups: "GD with Insulin treatment" versus "GD without Insulin treatment" In each group, the serum fructosamines rate will be estimated with a confidence interval of 95% and compared from a Student test.
  Interventions: Other: Fructosamines
- GD without Insulin treatment (Other): At the end of the study patients will be divided into two groups: "GD with Insulin treatment" versus "GD without Insulin treatment" In each group, the serum fructosamines rate will be estimated with a confidence interval of 95% and compared from a Student test.
  Interventions: Other: Fructosamines

INTERVENTIONS:
Other: Fructosamines

SUMMARY:
The prevalence of gestational diabetes is estimated at between 2 and 6%, but can be much higher in specific populations.

The specific treatment of gestational diabetes (diet, control weight gain, self monitoring glucose , insulin therapy) reduces complications severe perinatal, fetal macrosomia, and preeclampsia compared with abstention therapy, without additional risk of caesarean section.

Several early studies have shown that the determination of fructosamine is a very bad way of diagnosis for Gestational Diabetes. However, few studies have investigated the relationship between the determination of serum fructosamine and put under insulin in case of Gestational Diabetes.

The purpose of this study is to determine if serum fructosamines rate can be a predictive marker of the starting insulin at the patients suffering from Gestational Diabetes

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ongoing pregnancy with a start date of pregnancy known and confirmed by an ultrasound of the 1st Quarter performed between 10 and 14 weeks with measurement of the crown-rump length
* Hospitalization for a GD's discovery whatever the term of pregnancy (GD is defined with nationals recommendations of CNGOF)
* Not opposed to participate in the study

Exclusion Criteria:

* Pregnancy uncertain term (absence of early ultrasound)
* Previous diabetes to the pregnancy (type 1 or 2)
* Multiple Pregnancy
* No affiliation to a social security scheme
* Woman with a measure of legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Serum fructosamine rate | at baseline (when gestational diabetes is diagnosed: between 24 and 28 weeks of gestation or later)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DUCARME, PH, Principal Investigator — Centre Hospitalier Départemental Vendée
Locations (1):
- Centre hospitalier départemental Vendée, La Roche-sur-Yon, France

REFERENCES:
- [Background] Ducarme G, Desroys Du Roure F, Le Thuaut A, Grange J, Dimet J, Crepin-Delcourt I. Efficacy of maternal and biological parameters at the time of diagnosis of gestational diabetes mellitus in predicting neonatal morbidity. Eur J Obstet Gynecol Reprod Biol. 2018 Feb;221:113-118. doi: 10.1016/j.ejogrb.2017.12.036. Epub 2017 Dec 19. PMID 29278829
- [Result] Ducarme G, Desroys du Roure F, Grange J, Vital M, Le Thuaut A, Crespin-Delcourt I. Predictive factors of subsequent insulin requirement for glycemic control during pregnancy at diagnosis of gestational diabetes mellitus. Int J Gynaecol Obstet. 2019 Mar;144(3):265-270. doi: 10.1002/ijgo.12753. Epub 2019 Jan 11. PMID 30578686